CLINICAL TRIAL: NCT03628053
Title: Tisagenlecleucel Versus Blinatumomab or Inotuzumab for Adult Patients With Relapsed/Refractory B-cell Precursor Acute Lymphoblastic Leukemia: A Randomized Open Label, Multicenter, Phase III Trial
Brief Title: Tisagenlecleucel vs Blinatumomab or Inotuzumab for Patients With Relapsed/Refractory B-cell Precursor Acute Lymphoblastic Leukemia
Acronym: OBERON
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Novartis is no longer pursuing this study because of planned investigation of novel CAR-T therapies in this patient population.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019I2301
Record Dates: First submitted 2018-06-28; First posted 2018-08-14 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute lymphoblastic leukemia; tisagenlecleucel; intouzumab; blinatumomab; CAR-T; CTL019
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — tisagenlecleucel; blinatumomab; Inotuzumab Ozogamicin

STUDY DESIGN:
Intervention Model Description: This is a phase III, open label, multinational, randomized trial. Eligible patients will be randomized 1:1 to Tisagenlecleucel treatment strategy (tisagenlecleucel after optional bridging chemotherapy and lymphodepleting chemotherapy) or control arm treatment strategy (blinatumomab or inotuzumab per investigator's discretion after optional bridging chemotherapy).
  The randomization will be performed stratifying for the number of prior salvage therapies (0 vs. 1) and prior allogenic stem cell transplant (yes vs. no).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tisagenlecleucel arm (Experimental): Patient to receive tisagenlecleucel after optional bridging therapy and lymphodepleting chemotherapy.
  Interventions: Biological: Tisagenlecleucel
- Control arm (Active Comparator): blinatumomab or inotuzumab per investigator's discretion after optional bridging chemotherapy
  Interventions: Drug: Blinatumomab; Drug: Inotuzumab

INTERVENTIONS:
Biological: Tisagenlecleucel — autologous cellular immunotherapy product
  Other Names: CTL019; KYMRIAH
  Arms: Tisagenlecleucel arm
Drug: Blinatumomab — bispecific CD19-directed CD3 T-cell engager
  Other Names: BLINCYTO
  Arms: Control arm
Drug: Inotuzumab — CD22-directed antibody-drug conjugate
  Other Names: BESPONSA; Inotuzumab ozogamicin
  Arms: Control arm

SUMMARY:
This trial aims to compare the benefits and risks of tisagenlecleucel to blinatumomab or inotuzumab in adult patients with relapsed or refractory ALL. This trial investigates tisagenlecleucel as an additional treatment option for this patient population with high unmet medical need.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Age ≥ 18 years.
3. Subject with CD19-expressing B-ALL.
4. Adequate organ function.
5. Patients considered in any of the following settings are eligible:

   1. Untreated first or second relapse
   2. Refractory to primary induction therapy
   3. Refractory to first salvage therapy or
   4. Relapse after allogenic stem cell transplant.

Exclusion Criteria:

1. Patients presenting with untreated first relapse of ALL more than 24 months after initial diagnosis
2. Presence of extra-medullary disease.
3. History or presence of clinically relevant CNS pathology, or uncontrolled CNS leukemia.
4. History of Veno-occlusive Disease (VOD).
5. Active neurological autoimmune or inflammatory disorders.
6. Active acute Graft-versus-Host Disease (GvHD), grade 2-4.

Other protocol-defined Inclusion/Exclusion may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-05 (Estimated); Primary Completion 2025-10-08 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 4 years
  Time from randomization to death for any reason

SECONDARY OUTCOMES:
Event Free Survival (EFS) | 4 years
  EFS, assessed up to 48 months, is defined as the date from randomization to the earliest of (a) date of death due to any cause, (b) relapse after CR/CRi, or (c) treatment failure, which is defined as failure to achieve remission within 12 weeks of randomization.
Percentage of patients who achieved MRD negative CR/CRi | 4 years
  Percentage of patients who achieved MRD negative CR/CRi at month 3 post randomization
Overall response rate | 4 years
  ORR is defined as the proportion of subjects with best overall response (BOR) of CR or CRi, where the BOR is defined as the best response recorded from randomization until the start of new anticancer therapy or the data cut-off date, whichever is earlier
Duration of response (DOR) | 4 years
  DOR is defined as the duration from the date when the response criteria of CR/CRi is first met to the date of relapse or death due to underlying cancer.
Probability of patients who achieved CR/CRi at month 12 | 4 years
  Probability of achieving CR/CRi based on all response assessments between randomization and month 12. This outcome measure will be based on all randomized patients and the assessment will be up to 48 months (from randomization of the first patient until 12 months after the randomization of the last patient).
Prevalence of immunogenecity | 4 years
  Percentage of patients who have anti-tisagenlecleucel antibodies in the serum before randomization
Incidence of immunogenecity | 4 years
  Percentage of patients who develop anti-tisagenlecleucel antibodies in the serum after infusion of tisagenlecleucel
Impact of immunogenicity on clinical response | 4 years
  difference in response between patients with immunogenicity and patients without immunogenicity
Cellular kinetic profile by qPCR | 4 years
  Summary of qPCR detected tisagenlecleucel transgene concentrations
Cellular kinetics profile by flow cytometry | 4 years
  Summary of flow cytometry-detected tisagenlecleucel transgene concentrations
Relationship between dose and response | 4 years
  Relationship between the administered dose of tisagenlecleucel and response to treatment (complete response with or without hematological recovery). This assessment will be done for all patients for up to 48 months.
Relationship between exposure and response | 4 years
  Describe the relationship between the cellular kinetics of tisagenlecleucel overtime and response.
Relationship between dose and cellular kinetic | 4 years
  Describe the relationship between the dose of tisagenlecleucel actually administered and cellular kinetics
EQ-5D-3L | 4 years
  Patient reported outcome measure
EORTC QLQ-30 | 4 years
  Patient reported outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com